CLINICAL TRIAL: NCT06178094
Title: The Effects of Video Training Given to Individuals With Type 2 Diabetes Through Smartphones on Self-Care and Metabolic Control
Brief Title: The Effects of Video Training Given to Individuals With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, İlknur METİN AKTEN, assistant professor, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-69456409-199-35238
Record Dates: First submitted 2023-10-30; First posted 2023-12-20 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus, Type 2; Training
Keywords: Diabetes training,; Metabolic control variables; Self-care; Type 2 Diabetes; Video training
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Diabetes Training group (Experimental): The data collection tools will apply in the first and second interviews and metabolic control variables will record.
  Diabetes training videos will sent to the Training Group through smartphones after the first meeting as two episodes a week.
  Interventions: Behavioral: Video Training
- control group (No Intervention): The data collection tools will apply in the first and second interviews and metabolic control variables will record.

INTERVENTIONS:
Behavioral: Video Training — The participants in the Training Group is to sent a total of eight episodes of the Diabetes Training Videos prepare by the researcher, twice a week, through smartphones after the first interview
  Arms: Video Diabetes Training group

SUMMARY:
The goal of this randomised control type of study is to examine the effects of Video Diabetes Training given to individuals with Type 2 Diabetes through smartphones on self-care and metabolic control.

The Hypotheses of the Study:

H1: Video Diabetes Training given to individuals with Type 2 Diabetes through smartphones has a positive impact on individuals' self-care.

H2: Video Diabetes Training given to individuals with Type 2 Diabetes through smartphones has a positive impact on individuals' metabolic control variables.

Participants will answer the data collection tools in the first and second interviews and metabolic control variables will be record. Diabetes training videos will sent to the Training Group through smartphones after the first meeting as two episodes a week.

Video Diabetes Training given to training group will be examine the effects of on self-care and metabolic control.

DETAILED DESCRIPTION:
The study will conduct to examine the effects of Video Diabetes Training given to individuals with Type 2 Diabetes through smartphones on self-care and metabolic control.

This experimental, randomized, and controlled study will conduct with a total of 112 individuals with Type 2 Diabetes (56 in the Training Group, and 56 in the Control Group), who apply to the Internal Medicine Clinic of a state hospital in the Mediterranean Region of Turkey between February and August 2022, who volunteered to participate in the study and met the inclusion criteria.

A total of 112 individuals with Type 2 Diabetes, who volunteered to participate in the study, and met the inclusion criteria, will select with the Simple Random Sampling Method and will randomize with the help of a computer program.

Participants will answer the data collection tools in the first and second interviews and metabolic control variables will be record. Diabetes training videos will sent to the Training Group through smartphones after the first meeting as two episodes a week.

Video Diabetes Training given to training group will be examine the effects of on self-care and metabolic control.

ELIGIBILITY:
Inclusion Criteria:

* agreed to participate in the study voluntarily,
* were diagnosed with Type 2 Diabetes for at least 6 months,
* were 18 years of age or older,
* were literate, had smartphones with video playback features and internet,
* without a physician diagnosis that would prevent communication, and psychiatric problems and hearing problems
* those who did not have sensory losses such as vision or hearing.

Exclusion Criteria:

-Individuals who did not meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Numerical distribution of participants' sociodemographic and diabetes-related characteristics | At the first meeting (initial)
  The sociodemographic and diabetes-related characteristics of the training and control groups.
  Sociodemographic characteristics; Age, gender, marital status, education level, occupation, income level, smoking and alcohol use were evaluated.
  Characteristics of diabetes: duration of diabetes, diabetes treatment method, use of other medications, family history of diabetes, frequency of check-ups, hospitalization due to high blood sugar, hospitalization due to hypoglycemia, chronic complications due to diabetes, previous education on diabetes, status other than diabetes the presence of the disease was evaluated.
Diabetes Self-Care Scale mean score | At the first interview (baseline) and at the second interview 3 months later
  The comparison of Diabetes Self-Care Scale pre-test, post-test and change difference values between training and control groups. The lowest acceptable level of the scale is 92 points. The highest score that can be obtained from the scale is 140 points. As the score of the scale increases, patients' self-care activities also increase positively.
Fasting plasma glucose value | At the first interview (baseline) and at the second interview 3 months later
  Comparison of fasting plasma glucose variables between training and control groups.
  Fasting plasma glucose (mg/dl) value was obtained as a result of the participant's routine blood test.
HbA1c value | At the first interview (baseline) and at the second interview 3 months later
  Comparison of HbA1c variables between training and control groups. HbA1c (%) value was obtained as a result of the participant's routine blood test.
Total cholesterol value | At the first interview (baseline) and at the second interview 3 months later
  Comparison of total cholesterol variables between training and control groups. Total cholesterol (mg/dl) value was obtained as a result of the participant's routine blood test.
Low-density lipoprotein value | At the first interview (baseline) and at the second interview 3 months later
  Comparison of low-density lipoprotein variables between training and control groups.
  Low density lipoprotein (mg/dl) value was obtained as a result of the participant's routine blood test.
High-density lipoprotein value | At the first interview (baseline) and at the second interview 3 months later
  Comparison of high-density lipoprotein variables between training and control groups.
  High density lipoprotein (mg/dl) value was obtained as a result of the participant's routine blood test.
Triglyceride value | At the first interview (baseline) and at the second interview 3 months later
  Comparison of triglyceride variables between training and control groups. Triglyceride (mg/dl) value was obtained as a result of the participant's routine blood test.
Systolic blood pressure value | At the first interview (baseline) and at the second interview 3 months later
  Comparison of systolic blood pressure (mmHg) variables between training and control groups.
  The tools required for blood pressure measurement were provided by the researcher. The same measurement tools were used in the first interview (pretest) and the second interview (posttest). The participant was allowed to rest for at least 5-10 minutes before the measurement. An aneroid type sphygmomanometer, suitable for adults, was used as a measurement tool. In accordance with the technique recommended in the National Hypertension Treatment and Follow-up Guide, the researcher took measurements twice with an interval of two minutes while the participant was in a sitting position, with his right arm supported at heart level, and the results were recorded by averaging the measurements.
Diastolic blood pressure value | At the first interview (baseline) and at the second interview 3 months later
  Comparison of diastolic blood pressure (mmHg) variables between training and control groups.
  The tools required for blood pressure measurement were provided by the researcher. The same measurement tools were used in the first interview (pretest) and the second interview (posttest). The participant was allowed to rest for at least 5-10 minutes before the measurement. An aneroid type sphygmomanometer, suitable for adults, was used as a measurement tool. In accordance with the technique recommended in the National Hypertension Treatment and Follow-up Guide, the researcher took measurements twice with an interval of two minutes while the participant was in a sitting position, with his right arm supported at heart level, and the results were recorded by averaging the measurements.
Body Mass Index value | At the first interview (baseline) and at the second interview 3 months later
  Comparison of body mass index variables between training and control groups. To calculate the body mass index of the participants, they were measured according to the weight and height technique. Participants' BMI was calculated by dividing their weight by the square of their height [BMI: Weight (kg)/height (m2)]. BMI was evaluated in accordance with WHO recommendations.
Waist circumference value | At the first interview (baseline) and at the second interview 3 months later
  Comparison of waist circumference variables between training and control groups.
  Waist circumference measurement was made using the measurement technique recommended by WHO. While the participants were standing, the circumference was measured with a tape measure over their underwear, at the midpoint between the lowest rib and the crista iliaca at the end of expiration.

CONTACTS AND LOCATIONS:
Overall Officials: İlknur METİN AKTEN, PhD,MSc,RN, Principal Investigator — Kırklareli University
Locations (1):
- Kırklareli University, Kırklareli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kang J, Chen Y, Zhao Y, Zhang C. Effect of remote management on comprehensive management of diabetes mellitus during the COVID-19 epidemic. Prim Care Diabetes. 2021 Jun;15(3):417-423. doi: 10.1016/j.pcd.2020.12.004. Epub 2021 Jan 1. PMID 33422431
- [Result] Hansen CR, Perrild H, Koefoed BG, Zander M. Video consultations as add-on to standard care among patients with type 2 diabetes not responding to standard regimens: a randomized controlled trial. Eur J Endocrinol. 2017 Jun;176(6):727-736. doi: 10.1530/EJE-16-0811. Epub 2017 Mar 21. PMID 28325823
- [Result] Lee NP, Fisher WP Jr. Evaluation of the Diabetes Self-Care Scale. J Appl Meas. 2005;6(4):366-81. PMID 16192661
- [Result] Avdal EU, Uran BNO, Pamuk G, Yildirim JG, Konakci G, Ates M, Polat G. Investigation of the effect of web-based diabetes education on metabolic parameters in people with type 2 diabetes: A randomized controlled trial. J Infect Public Health. 2020 Dec;13(12):1892-1898. doi: 10.1016/j.jiph.2020.03.008. Epub 2020 May 20. PMID 32444190
- [Result] Bell AM, Fonda SJ, Walker MS, Schmidt V, Vigersky RA. Mobile phone-based video messages for diabetes self-care support. J Diabetes Sci Technol. 2012 Mar 1;6(2):310-9. doi: 10.1177/193229681200600214. PMID 22538140
- [Result] Rasmussen OW, Lauszus FF, Loekke M. Telemedicine compared with standard care in type 2 diabetes mellitus: A randomized trial in an outpatient clinic. J Telemed Telecare. 2016 Sep;22(6):363-8. doi: 10.1177/1357633X15608984. Epub 2015 Oct 14. PMID 26468213
- [Result] Sun C, Sun L, Xi S, Zhang H, Wang H, Feng Y, Deng Y, Wang H, Xiao X, Wang G, Gao Y, Wang G. Mobile Phone-Based Telemedicine Practice in Older Chinese Patients with Type 2 Diabetes Mellitus: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Jan 4;7(1):e10664. doi: 10.2196/10664. PMID 30609983
- [Result] Tang PC, Overhage JM, Chan AS, Brown NL, Aghighi B, Entwistle MP, Hui SL, Hyde SM, Klieman LH, Mitchell CJ, Perkins AJ, Qureshi LS, Waltimyer TA, Winters LJ, Young CY. Online disease management of diabetes: engaging and motivating patients online with enhanced resources-diabetes (EMPOWER-D), a randomized controlled trial. J Am Med Inform Assoc. 2013 May 1;20(3):526-34. doi: 10.1136/amiajnl-2012-001263. Epub 2012 Nov 20. PMID 23171659